CLINICAL TRIAL: NCT03898154
Title: The Effect on Wrist Range of Motion With Perioperative Glucocorticoid Administration in the Treatment of Adult Distal Radius Fractures: A Randomized Controlled Trial
Brief Title: Perioperative Glucocorticoid Administration in the Treatment of Adult Distal Radius Fractures
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: C. Liam Dwyer (Other)
Responsible Party: Sponsor-Investigator, C. Liam Dwyer, Staff Physician, Geisinger Clinic
Organization: Geisinger Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0533
Record Dates: First submitted 2019-03-28; First posted 2019-04-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures | interventions — Dexamethasone; Methylprednisolone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Glucocorticoid (GC) group (Experimental): Intraoperative: Single intraoperative dose of 10 mg intravenous dexamethasone Postoperative: A 6-day oral methylprednisolone (oral GC) taper course. The oral GC taper course begins on the day of surgery and includes 24mg on day 1, 20mg on day 2, 16mg on day 3, 12mg on day 4, 8mg on day 5, and 4mg on day 6
  Interventions: Drug: Dexamethasone; Drug: Methylprednisolone
- Control (non-GC) group (No Intervention): No GC administration

INTERVENTIONS:
Drug: Dexamethasone — Intraoperative: Single intraoperative dose of 10 mg intravenous dexamethasone
  Arms: Glucocorticoid (GC) group
Drug: Methylprednisolone — Postoperative: A 6-day oral methylprednisolone (oral GC) taper course. The oral GC taper course begins on the day of surgery and includes 24mg on day 1, 20mg on day 2, 16mg on day 3, 12mg on day 4, 8mg on day 5, and 4mg on day 6
  Arms: Glucocorticoid (GC) group

SUMMARY:
The purpose of this investigation is to compare functional outcome measures and range of motion for patients receiving glucocorticoid (GC) injections versus those not receiving GCs for the treatment of distal radius fractures. The investigators hypothesize that patients who receive GC will have improved ROM and functional outcome measures compared to patients who do not receive GC. In addition, this study aims to determine if there is a difference in rates of complications and postoperative pain control between the GC and non-GC groups. In order to accomplish these aims, the investigators will conduct a prospective, randomized, controlled investigation.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age and older.
* Patients undergoing ORIF with VP fixation of an acute, isolated DRF with or without associated distal ulna fracture and with or without associated carpal tunnel release

Exclusion Criteria:

* Worker's compensation patient
* Non-operatively treated fractures
* Open fractures
* Preoperative neurovascular injury
* Coexisting fractures or injuries
* Diabetes mellitus
* Allergy or contraindication to GCs
* Associated non-orthopedic injury that would prohibit the administration of GCs
* Patients currently incarcerated
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-07-10 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
QuickDASH | 0-12 months
  best 0-100 worst; functional outcome score for disabilities of the arm, shoulder, and hand
Visual Analog Scale Pain Score | 0-12 months
  best 0-10 worst; continuous scale to measure current pain level
PROMIS Pain Interference | 0-12 months
  best 0-100 worst; measures the effects of a patient's pain on their daily activities and lifestyle
PROMIS Self-Efficacy Manage Symptoms | 0-12 months
  best 0-100 worst; measures a patient's ability to cope with their symptoms related to the procedure
PROMIS Upper Extremity | 0-12 months
  worst 0-100 best; measures physical function of upper extremities

CONTACTS AND LOCATIONS:
Overall Officials: Liam Dwyer, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Woodbine, Danville, Pennsylvania, United States